CLINICAL TRIAL: NCT00597350
Title: Pilot Study of the Effect of Fenugreek on Blood Sugar and Insulin in Diabetic Humans
Brief Title: Effect of Fenugreek on Blood Sugar and Insulin in Diabetic Humans
Acronym: Fenugreek
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Frank Greenway, Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 27031
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus
Keywords: Fenugreek; Trigonella foenum-graecum; Diabetes mellitus; Blood sugar; Insulin; Glucose
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — fenugreek seed meal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood drawn for glucose and insulin levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Group with diabetes mellitus
  Interventions: Dietary Supplement: Trigonella foenum-graecum (fenugreek)

INTERVENTIONS:
Dietary Supplement: Trigonella foenum-graecum (fenugreek) — 2 slices of bread containing 5 grams of the natural herb fenugreek 2 times, 1 week apart

SUMMARY:
The purpose of this study is to determine if bread containing fenugreek reduces blood sugar and insulin compared to identical bread without fenugreek.

DETAILED DESCRIPTION:
Trigonella foenum-graecum (fenugreek) has been used in traditional medicine for the treatment of diabetes. Fenugreek has been demonstrated to lower blood glucose in response to a glucose load while leaving the levels of serum insulin unaffected in rodents. This effect of lowering blood sugar without changing insulin levels demonstrates improved insulin action. Fenugreek has also been shown to decrease glucose absorption by inhibiting intestinal disaccharidases. Fenugreek decreases glycohemoglobin in diabetic rodents. An amino acid extracted from fenugreek seeds, 4-hydroxyisoleucine, decreases glucose and insulin in diabetic rodents, improves glucose tolerance and stimulates insulin secretion from isolated pancreatic rodent islets.

Fenugreek imparts a bitter taste to products into which it is placed, and this property has limited its use in treating diabetes. Dr. Losso and his associates developed a process that allows incorporation of fenugreek into bread and other bakery goods without imparting a bitter taste, and the success of this process was confirmed in taste testing. This study is designed to evaluate the effect of fenugreek bread made by Dr. Losso's proprietary process on glucose and insulin.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female with diet controlled diabetes mellitus.
* Between 18 and 70 years of age.

Exclusion criteria:

* Pregnant or nursing.
* Taking medication for diabetes or a medication like oral cortisone that is known to affect blood sugar or blood insulin.
* Taking any chronic medication that has not had a stable dose for 1 month or longer. Oral contraceptives are accepted.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Area under the curve for insulin and glucose | 4 hrs. after eating the bread

SECONDARY OUTCOMES:
Any adverse event experienced by the subjects | 2 times, 1 wk. apart

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, M.D., Principal Investigator — Pennington Biomedical Research Center; Amber Torres, RD, LDN, Study Director — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Hannan JM, Ali L, Rokeya B, Khaleque J, Akhter M, Flatt PR, Abdel-Wahab YH. Soluble dietary fibre fraction of Trigonella foenum-graecum (fenugreek) seed improves glucose homeostasis in animal models of type 1 and type 2 diabetes by delaying carbohydrate digestion and absorption, and enhancing insulin action. Br J Nutr. 2007 Mar;97(3):514-21. doi: 10.1017/S0007114507657869. PMID 17313713
- [Background] Xue WL, Li XS, Zhang J, Liu YH, Wang ZL, Zhang RJ. Effect of Trigonella foenum-graecum (fenugreek) extract on blood glucose, blood lipid and hemorheological properties in streptozotocin-induced diabetic rats. Asia Pac J Clin Nutr. 2007;16 Suppl 1:422-6. PMID 17392143
- [Background] Broca C, Gross R, Petit P, Sauvaire Y, Manteghetti M, Tournier M, Masiello P, Gomis R, Ribes G. 4-Hydroxyisoleucine: experimental evidence of its insulinotropic and antidiabetic properties. Am J Physiol. 1999 Oct;277(4):E617-23. doi: 10.1152/ajpendo.1999.277.4.E617. PMID 10516120